CLINICAL TRIAL: NCT01707472
Title: A Phase 2a Study of an Anti-LOXL2 Monoclonal Antibody (GS-6624) in HIV and/or Hepatitis C- Infected Subjects With Liver Fibrosis
Brief Title: Study of Simtuzumab in HIV and/or Hepatitis C- Infected Adults With Liver Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-321-0107
Record Dates: First submitted 2012-09-11; First posted 2012-10-16 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Liver Fibrosis; Hepatitis C; HIV; HIV/HCV Co-infection
Keywords: Liver Fibrosis; Fibrosis; HIV; HCV; GS-6624; Hepatitis; Hepatitis C
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C; Fibrosis; Hepatitis | interventions — simtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Simtuzumab in HIV Patients (Experimental): HIV-infected participants will receive simtuzumab every 2 weeks for 24 weeks while continuing on standard therapy for HIV.
  Interventions: Biological: Simtuzumab
- Simtuzumab in HCV Patients (Experimental): HCV-infected participants will receive simtuzumab every 2 weeks for 24 weeks.
  Interventions: Biological: Simtuzumab
- Simtuzumab in HIV/HCV Co-Infected Patients (Experimental): HIV/HCV co-infected participants will receive simtuzumab every 2 weeks for 24 weeks while continuing on standard therapy for HIV.
  Interventions: Biological: Simtuzumab

INTERVENTIONS:
Biological: Simtuzumab — 700 mg intravenously for a total of 12 infusions.
  Other Names: Anti-LOXL2 Monoclonal Antibody; GS-6624

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of simtuzumab (formerly GS-6624) in HIV and/or hepatitis C virus (HCV)-infected adults with evidence of liver fibrosis.

ELIGIBILITY:
Key Inclusion Criteria:

* HIV-infected individuals must have positive serologies with viral load suppressed below 400 copies/mL
* HCV-infected individuals must have:

  * Chronic HCV infection with HCV RNA ≥ 2000 IU/ml AND at least 1 of the following:
  * Been null responder to previous pegylated interferon and ribavirin therapy OR
  * Failed to achieve sustained virologic response (SVR) on a regimen containing a direct-acting antiviral (DAA) in addition to pegylated interferon and ribavirin OR
  * Are unwilling to receive or have contraindications to interferon therapy for HCV
* HIV/HCV co-infected individuals must have:

  * Positive HIV serologies with viral load suppressed below 400 copies/mL
  * Chronic HCV infection with HCV RNA ≥ 2000 IU/ml AND at least 1 of the following:
  * Been null responder to previous pegylated interferon and ribavirin therapy OR
  * Failed to achieve SVR on a regimen containing a direct-acting antiviral (DAA) in addition to pegylated interferon and ribavirin OR
  * Are unwilling to receive or have contraindications to interferon therapy for HCV
* Willing to allow blood and tissue samples to be stored for future use to study HIV infection, immune function, liver disease and additional mechanisms involved in liver fibrosis among patients with HIV and/or HCV, which may not be related directly to the specific objectives of this study protocol
* Have a primary care physician

Key Exclusion Criteria:

* Cause of liver fibrosis other than HCV or long-term antiretroviral therapy (ART) treatment for HIV
* Currently being treated for HCV
* Evidence of active Hepatitis A, B or D infections
* History or evidence of hepatocellular carcinoma
* Unwillingness to undergo a liver biopsy pre-treatment and post-treatment, or to undergo all other protocol required tests/procedures or return to the site for required visits
* Presence of contraindications to magnetic resonance imaging (e.g., presence of any metal in the body, cardiac or neural pacemaker, aneurysm clip, cochlear implant, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2014-10-17 (Actual); Study Completion 2014-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- NIH Department of Laboratory Medicine, Bethesda, Maryland, United States

REFERENCES:
- [Background] Meissner EG, McLaughlin M, Matthews LA, Kanwar B, Bornstein JD, Kovacs JA, et al. Longitudinal hepatic and PBMC gene expression profiling of HIV and/or HCV-infected patients with advanced liver disease treated with simtuzumab, an anti-LOXL2 antibody [Abstract 448]. Hepatology AASLD Abstracts 2014;60 Number 4 (Suppl):421A.
- [Background] Han MAT, Gharib AM, Zhao X, Sinkus R, Rizvi BS, Matthews L, et al. Noninvasive Measures of Severity in Chronic Liver Disease, Moving Beyond Fibrosis [Abstract Sa1006]. Digestive Disease Week; 2015 16-19 May; Washington, D.C.
- [Derived] Gharib AM, Han MAT, Meissner EG, Kleiner DE, Zhao X, McLaughlin M, Matthews L, Rizvi B, Abd-Elmoniem KZ, Sinkus R, Levy E, Koh C, Myers RP, Subramanian GM, Kottilil S, Heller T, Kovacs JA, Morse CG. Magnetic Resonance Elastography Shear Wave Velocity Correlates with Liver Fibrosis and Hepatic Venous Pressure Gradient in Adults with Advanced Liver Disease. Biomed Res Int. 2017;2017:2067479. doi: 10.1155/2017/2067479. Epub 2017 Apr 5. PMID 28480218
- [Derived] Meissner EG, McLaughlin M, Matthews L, Gharib AM, Wood BJ, Levy E, Sinkus R, Virtaneva K, Sturdevant D, Martens C, Porcella SF, Goodman ZD, Kanwar B, Myers RP, Subramanian M, Hadigan C, Masur H, Kleiner DE, Heller T, Kottilil S, Kovacs JA, Morse CG. Simtuzumab treatment of advanced liver fibrosis in HIV and HCV-infected adults: results of a 6-month open-label safety trial. Liver Int. 2016 Dec;36(12):1783-1792. doi: 10.1111/liv.13177. Epub 2016 Jul 6. PMID 27232579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 04 October 2012. The last study visit occurred on 17 October 2014.
Pre-assignment Details: 37 participants were screened.
Groups:
- Simtuzumab in HIV Participants: Participants with human immunodeficiency virus (HIV) received simtuzumab 700 mg intravenously every 2 weeks over a period of 24 weeks while continuing on standard therapy for HIV.
- Simtuzumab in HCV Participants: Participants with hepatitis C virus (HCV) received simtuzumab 700 mg intravenously every 2 weeks over a period of 24 weeks.
- Simtuzumab in HIV/HCV Co-Infected Participants: Participants co-infected with HIV and HCV received simtuzumab 700 mg intravenously every 2 weeks over a period of 24 weeks while continuing on standard therapy for HIV.
Period: Overall Study
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Started | 4 | 6 | 8
Completed | 4 | 6 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least one dose of study drug.
Groups:
- Simtuzumab in HIV Participants: Participants with HIV received simtuzumab 700 mg intravenously every 2 weeks over a period of 24 weeks while continuing on standard therapy for HIV.
- Simtuzumab in HCV Participants: Participants with HCV received simtuzumab 700 mg intravenously every 2 weeks over a period of 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants | Total
Number analyzed (Participants) | 4 | 6 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (6.3) | 58 (5.0) | 54 (5.6) | 56 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 4
  Male | 4 | 3 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 6 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 2 | 4 | 6
  White | 2 | 4 | 2 | 8
  American Indian or Alaska native | 0 | 0 | 1 | 1
  Other | 2 | 0 | 1 | 3
Ishak Fibrosis Score [Count of Participants; unit: Participants] — The Ishak fibrosis score measures the degree of liver fibrosis (scarring) and ranges from 0 (best) to 6 (worst).
  Participants
    Stage 0 | 0 | 0 | 0 | 0
    Stage 1 | 0 | 0 | 0 | 0
    Stage 2 | 0 | 0 | 0 | 0
    Stage 3 | 1 | 1 | 4 | 6
    Stage 4 | 1 | 0 | 1 | 2
    Stage 5 | 0 | 1 | 1 | 2
    Stage 6 | 2 | 4 | 2 | 8
Hepatic Venous Pressure Gradient (HVPG) [Mean (Standard Deviation); unit: millimeters of Mercury (mm Hg)] | 8 (5.3) | 9 (3.7) | 8 (3.7) | 8 (3.8)
Morphometric Quantitative Collagen (MQC) [Mean (Standard Deviation); unit: percentage of MQC] | 4.24 (2.414) | 11.79 (9.582) | 12.75 (14.596) | 10.54 (11.312)
Alpha Smooth Muscle Actin (alpha SMA) [Mean (Standard Deviation); unit: percentage of alpha-SMA] | 6.59 (4.351) | 12.58 (12.184) | 13.32 (15.803) | 11.58 (12.549)
Magnetic Resonance Elastography (MRE) [Mean (Standard Deviation); unit: kPa] — Liver fibrosis is measured by MRE in kilopascal (kPa)
  kPa | 2.19 (0.370) | 2.01 (0.322) | 2.32 (0.487) | 2.20 (0.399)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: First dose date up to Week 24 plus 30 days
Population: The Safety Analysis Set included participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Number analyzed (Participants) | 4 | 6 | 8
percentage of participants | 100 | 100 | 100

2. Secondary Outcome: Number of Participants With a Change From Baseline in Ishak Fibrosis Stage Score at Week 24
Description: The Ishak fibrosis score measures the degree of liver fibrosis (scarring) and ranges from 0 (best) to 6 (worst). A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set (who were enrolled into the study and received at least 1 dose of study drug) with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Number analyzed (Participants) | 3 | 6 | 8
Participants
  Fibrosis improved: -2 | 0 | 1 | 0
  Fibrosis improved: -1 | 1 | 1 | 0
  Fibrosis did not change: 0 | 2 | 4 | 5
  Fibrosis worsened: 1 | 0 | 0 | 2
  Fibrosis worsened: 2 | 0 | 0 | 1

3. Secondary Outcome: Change From Baseline in HVPG at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Number analyzed (Participants) | 4 | 6 | 8
mm Hg | 2 (2.4) | 0 (3.4) | 0 (1.1)

4. Secondary Outcome: Change From Baseline in MQC at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with liver biopsy area ≥ 4 mm^2 (adequate for morphometry measurements) were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of MQC
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Number analyzed (Participants) | 3 | 4 | 5
percentage of MQC | 2.07 (5.333) | -2.54 (11.510) | 1.27 (9.612)

5. Secondary Outcome: Change From Baseline in Alpha SMA at Week 24
Time Frame: Baseline; Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of alpha-SMA
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Number analyzed (Participants) | 3 | 4 | 5
percentage of alpha-SMA | 4.69 (3.938) | 5.27 (6.973) | 4.50 (7.669)

6. Secondary Outcome: Change From Baseline in Liver Fibrosis as Estimated by MRE at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
Number analyzed (Participants) | 4 | 3 | 5
kPa | 0.17 (0.141) | 0.09 (0.203) | 0.09 (0.085)

ADVERSE EVENTS:
Time Frame: First dose date to Week 24 plus 30 Days
Description: The Safety Analysis Set included participants who received at least one dose of study drug.
Arm/Group | Simtuzumab in HIV Participants | Simtuzumab in HCV Participants | Simtuzumab in HIV/HCV Co-Infected Participants
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 1/8
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simtuzumab in HIV Participants (N=4) | Simtuzumab in HCV Participants (N=6) | Simtuzumab in HIV/HCV Co-Infected Participants (N=8)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Gallbladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simtuzumab in HIV Participants (N=4) | Simtuzumab in HCV Participants (N=6) | Simtuzumab in HIV/HCV Co-Infected Participants (N=8)
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0
Infusion site rash (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 5 | 4
Amylase increased (Investigations) | 3 | 5 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 3
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 3
Blood bilirubin increased (Investigations) | 1 | 1 | 2
Blood creatine phosphokinase abnormal (Investigations) | 2 | 1 | 3
Blood creatinine decreased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 2
Blood lactate dehydrogenase abnormal (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 5 | 6
Haemoglobin decreased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 4 | 5
Lipase increased (Investigations) | 2 | 3 | 4
Platelet count decreased (Investigations) | 2 | 2 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 4 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years